CLINICAL TRIAL: NCT00005595
Title: Multicenter Phase II Trial of Arsenic Trioxide in Relapsed and Refractory Hodgkin's Disease
Brief Title: Arsenic Trioxide in Treating Patients With Relapsed or Refractory Hodgkin's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to accrue subjects in a timely fashion.
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NCI 99H5; NU-99H5; NCI-T99-0093
Record Dates: First submitted 2000-05-02; First posted 2004-03-04 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: arsenic trioxide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of arsenic trioxide in treating patients who have relapsed or refractory Hodgkin's disease.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of arsenic trioxide in terms of rate of response (complete or partial remission), duration of response, relapse free survival, and overall survival in patients with relapsed or refractory Hodgkin's disease. II. Evaluate the toxicities of this agent in this patient population. III. Elucidate the mechanism of action of this treatment by measuring induction of apoptosis and caspace activation when given to these patients.

OUTLINE: This is a multicenter study. Patients receive arsenic trioxide IV over 1-2 hours daily for up to 60 days. After 4-6 weeks of rest, patients receive up to 5 additional courses of therapy of 25 days each followed by 4-6 weeks of rest. Patients with a complete response (CR) receive 1 additional course of 25 days after achieving CR. Treatment continues in the absence of unacceptable toxicity or disease progression. Patients are followed monthly for 6 months, every 2 months for 6 months, every 3 months for 12 months, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 12-35 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed relapsed or refractory Hodgkin's disease Relapsed after prior first line treatment with at least 2 regimens, such as: Mechlorethamine, vincristine, procarbazine, and prednisone (MOPP) Doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) MOPP/ABV Stanford 5 OR Refractory to a second line regimen, such as: Mesna, ifosfamide, mitoxantrone, and etoposide (MINE) Etoposide, methylprednisolone, high dose cytarabine, and cisplatin (ESHAP) High dose chemotherapy and autologous or allogeneic stem cell transplantation At least 1 measurable lesion

PATIENT CHARACTERISTICS: Age: 16 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Unless documented bone marrow involvement: WBC at least 4,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2.0 mg/dL Renal: Creatinine no greater than 2.0 mg/dL Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception HIV negative No other prior malignancies within the past 5 years except curatively treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix No concurrent active infection requiring antibiotics

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics No concurrent biologic agents No concurrent monoclonal antibodies No concurrent bone marrow transplantation Chemotherapy: See Disease Characteristics No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No concurrent radiotherapy Surgery: Not specified Other: No other concurrent anticancer agents

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2000-06; Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin S. Tallman, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (2):
- United States (2):
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Memorial Sloan-Kettering Cancer Center, New York, New York